CLINICAL TRIAL: NCT02285335
Title: Effects of GINST on Human Semen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2014-0708
Record Dates: First submitted 2014-11-03; First posted 2014-11-07 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low group (Experimental): GINST15 3g/day
  Interventions: Dietary Supplement: GINST
- High group (Experimental): GINST15 6g/day
  Interventions: Dietary Supplement: GINST

INTERVENTIONS:
Dietary Supplement: GINST — The study is designed with using GINST either 500mg/capsule or 1000mg/capsule, two capsules at once, three times a day for 12 weeks.

SUMMARY:
The purpose of the study is to evaluate the effect of GINST on human semen. The study is a pilot study, designed as open-label, prospective randomized clinical trial using GINST either 500mg/capsule (panax ginseng 0.96g/day) or 1000mg/capsule (panax ginseng 1.92g/day), two capsules at once, three times a day for 12 weeks. GINST(Ilhwa, Republic of Korea) is a dietary supplement capsule, which is made with 6 year-old Korean red ginseng (Panax ginseng). Expected participants are to be male partners of female patients who visit infertility clinic at Severance hospital, whose total motile sperm count is more than 0.5x106 by semen analysis using computer aided sperm analyzer (CASA). Semen analysis, blood test, questionaires are planned to be performed 2 times, on the initial visit and after 12weeks of GINST treatment. Semen analysis will reveal ejaculated volume, sperm count, motility, morphology, total leukocyte count, total motile sperm count, further analysis including sperm chromatin assessment to examine the quality of sperm and malondialdehyde (MDA) analysis of seminal fluid to assess oxidative stress will be performed. Blood test will be done including serum follicle stimulating hormone (FSH), luteinizing hormone (LH), total and free testosterone. Quality of life, sexual performance before and after taking GINST will be evaluated using questionaires.

ELIGIBILITY:
Inclusion Criteria:

1. partner of female patient who visit infertility clinic with chief complaint of infertility.
2. ≥0.5x106 of total motile sperm count on screening semen analysis.

Exclusion Criteria:

1. Those who have chronic, systemic disease or endocrinologic disorder.
2. Patients with hypertension (systolic blood pressure ≥ 140mmHg, diastolic blood pressure ≥ 90mmHg)
3. Patients who have undergone chemotherapy due to malignancy
4. Patient who has history of taking testosterone or anti androgen agents within 1 month.
5. Patient who has retrieved sperm surgically

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Semen quality (assessed by computer aided semen analysis and sperm chromatin assay, malondialdehyde (MDA) analysis) | 12 week
  Semen quality assessed by computer aided semen analysis and sperm chromatin assay, malondialdehyde (MDA) analysis

SECONDARY OUTCOMES:
serum hormones (serum FSH(follicle stimulating hormone), LH(luteinizing hormone), testosterone) | 12 week
  serum FSH(follicle stimulating hormone), LH(luteinizing hormone), testosterone
Quality of Life (SF-36, Brief sexual function inventory, fatigue severity scale) | 12 week
  Assessment of quality of life by questionaire (SF-36, Brief sexual function inventory, fatigue severity scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea